CLINICAL TRIAL: NCT03446417
Title: A Phase 1/2 Open Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of ZN-e4 (KP-673) in Patients With Advanced Non-Small Cell Lung Cancer With Activating Epidermal Growth Factor Receptor (EGFR) Mutations
Brief Title: A Study of ZN-e4 in Subjects With Epidermal Growth Factor Receptor Mutated Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zeno Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZN-e4-001
Record Dates: First submitted 2018-02-16; First posted 2018-02-26 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Up to 9 sequential dose escalation cohorts to determine maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) is identified.
  Interventions: Drug: ZN-e4
- Phase 2 (Experimental): MTD/RP2D in subjects:
  Cohort 1: with T790M mutation in epidermal growth factor receptor (EGFR) gene, and are osimertinib naïve.
  Cohort 2: EGFRm amenable to EGFR inhibitor therapy (eg, exon 19 del, L858R) and who have never been treated with EGFRis.
  Interventions: Drug: ZN-e4

INTERVENTIONS:
Drug: ZN-e4 — Oral dose, tablet, daily dosing

SUMMARY:
This is a Phase 1/2, open-label, multicenter, sequential dose-escalation study to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of ZN-e4 administered orally in subjects with advanced non-small cell lung cancer (NSCLC) with activating EGFR mutations who have progressed while on treatment with an EGFR tyrosine kinase inhibitor (TKI) agent (other lines of treatment are allowed, except for other epidermal growth factor receptor inhibitors [EGFRis]) for Phase 1; and for Phase 2, subjects who have T790M+ and are osimertinib naïve (Cohort 1), and also those who have not been treated with an EGFR Inhibitor (EGFRi) (Cohort2).

ELIGIBILITY:
INCLUSION CRITERIA

* Age ≥ 18 years
* Histologically or cytologically confirmed metastatic or advanced inoperable diagnosis of NSCLC
* Documented radiographic progression on the last treatment administered prior to enrolling in the study.
* Phase 1 only: Confirmation that the tumor harbors an EGFR mutation known to be associated with aberrations that are amenable to EGFRi therapy including but not limited to: G719X, exon 19 deletion, exon 21 L858R, and L861Q. OR - Must have experienced clinical benefit from an EGFRi,
* All acute toxic effects of any prior antitumor therapy resolved to Grade ≤1 or baseline before the start of study drug dosing (with the exception of alopecia [any grade permitted] and neurotoxicity [Grade 1 or 2 permitted]).
* Measurable disease meeting the criteria specified by RECIST v1.1
* Phase 2, Cohort 1 only: Subjects must have confirmation of tumor T790M mutation status (confirmed positive) and are osimertinib naïve
* Phase 2, Cohort 2 only: EGFR aberrations that are amenable to EGFRi therapy, including but not limited to: G719X, exon 19 deletion, exon 21 L858R, and L861Q, and be EGFRi naïve

EXCLUSION CRITERIA

* Subjects who have received only neoadjuvant or adjuvant therapy for NSCLC.
* Phase 1 only: Treatment with an EGFRi within 7 days or 5 half-lives of the first dose of study treatment, whichever is shorter.
* Phase 1 only: Cytotoxic chemotherapy, investigational agents, or any anticancer therapy for the treatment of advanced NSCLC (other than EGFRi) within 21 days of the first dose of study treatment.
* Prior treatment with immunotherapy within 3 months prior to the first dose of study treatment.
* Radiotherapy within 28 days of first dose of study treatment; subjects given palliative radiotherapy to peripheral sites (e.g., bone metastases) may enter the study before 28 days have elapsed provided the radiated sites do not contain lesions which may be used to evaluate response, and must have recovered from any acute, reversible effects.
* Known or suspected central nervous system (CNS) metastases or leptomeningeal disease (Phase 1 only). Subjects with previously treated brain or CNS metastases are eligible provided that the subject has recovered from any acute effects of radiotherapy, does not have brain metastasis related symptoms, is not requiring systemic steroids for at least 2 weeks prior to study drug administration, and any whole brain radiation therapy was completed at least 4 weeks prior to study drug administration, or any stereotactic radiosurgery (SRS) was completed at least 2 weeks prior to study drug administration.
* Prior allogeneic bone marrow transplantation.
* History of a concurrent or second malignancy except for: adequately treated local basal cell or squamous cell carcinoma of the skin; cervical carcinoma in situ; superficial bladder cancer; breast carcinoma in situ; adequately treated Stage 1 or 2 cancer currently in complete remission; any other cancer that has been in complete remission for ≥5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Observed dose limiting toxicities | 1 Cycle (21 days)

SECONDARY OUTCOMES:
Safety and tolerability as measured by incidence of treatment emergent adverse events | Through study completion, approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zeno Pharmaceuticals, Study Director — Zeno Pharmaceuticals
Locations (7):
- United States (5):
  - Site 2, Duarte, California
  - Site 5, Detroit, Michigan
  - Site 1, East Setauket, New York
  - Site 6, Charlotte, North Carolina
  - Site 3, Gettysburg, Pennsylvania
- Bosnia and Herzegovina (2):
  - Site 8, Banja Luka
  - Site 7, Sarajevo

IPD SHARING:
Plan to Share IPD: No